CLINICAL TRIAL: NCT02277587
Title: A Randomized, Controlled, Multi-Centre Trial on the Effects of Dual-release Hydrocortisone Preparations Versus Conventional Glucocorticoid Replacement Therapy in Patients Affected by Primary and Secondary Adrenal Insufficiency. DREAM Trial.
Brief Title: Dual RElease Hydrocortisone Versus conventionAl Glucocorticoid replaceMent Therapy in Hypocortisolism (DREAM)
Acronym: DREAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyposurrenalism_1
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Primary Adrenal Insufficiency; Secondary Adrenal Insufficiency
Keywords: Plenadren; Addison's disease; Hydrocortisone; Cortisone Acetate; Monocytes; Natural Killer cells; Immunological profile; Inflammation
MeSH Terms: conditions — Addison Disease; Inflammation | interventions — Hydrocortisone; Cortisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Plenadren (Experimental): Plenadren (modified release hydrocortison) 20-25 or 30 mg oral tablets will be administered once-daily at 8.00 AM in the fasting state The dose is kept the same as patients had before entering the trial.
  Interventions: Drug: Plenadren
- Conventional glucocorticoid therapy (Active Comparator): Hydrocortisone (dose range 10 to 30) mg will be continued as before entering the study. Cortisone Acetate (dose 25 to 37.5 mg) will be continued as before entering the study. The morning dose will be administered in the fasting state.
  The total daily dose and timing is not changed during the study period.
  Interventions: Drug: Conventional glucocorticoid therapy
- Healthy volunteers (No Intervention): Healthy volunteers will be enrolled as control group

INTERVENTIONS:
Drug: Plenadren — Oral Tablets: 20-25-30 mg
  Other Names: Dual-release Hydrocortisone
  Arms: Plenadren
Drug: Conventional glucocorticoid therapy — Oral Tablets: 20-25-30- 37.5 mg
  Other Names: Hydrocortisone / Cortisone Acetate
  Arms: Conventional glucocorticoid therapy

SUMMARY:
This is a randomized, controlled, open, three-armed, multi-centre study designed to compare the effects of dual-release hydrocortisone preparations versus conventional glucocorticoid therapy on anthropometric parameters, metabolic syndrome, infectious, immunological profile, cardiovascular system, bone mass and quality of life in patients affected by primary or secondary adrenal insufficiency.

DETAILED DESCRIPTION:
Hypocortisolism is a disease with more than 80% 1-year mortality before the availability of synthetic glucocorticoids. Current replacement therapy has improved this dramatically, but recent data suggest that outcome is still compromised. Patient receiving conventional glucocorticoids therapy have compromised quality of life, reduced bone mass, increased risk factors for cardiovascular disease, infectious, tumors and premature mortality that is more than twice the mortality rate in the background population. Circulating cortisol levels follow a distinct diurnal pattern with high levels in the early morning and low trough values around midnight. Using available formulations for replacement therapy this circadian rhythm is had to mimic and also during the active time of the day high peaks and low troughs occur.

In this trial a dual-release hydrocortisone preparations that has in healthy volunteers been able to mimic the circadian pattern of circulating cortisol was studied in patients with primary and secondary adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed (e.g. more than 6 months ago) primary or secondary adrenal insufficiency with a stable daily glucocorticoid substitution dose for at least 3 months prior to study entry
* Signed informed consent to participate in the study

Exclusion Criteria:

* acute primary or secondary adrenal insufficiency
* clinical or laboratory signs of significant cerebral, cardiovascular, respiratory, hepatobiliary, pancreatic disease
* clinically significant renal dysfunction
* any medication with agents which could interfere with glucocorticoid kinetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in measurement of weight at 3 and 6 months | 0, + 3 months, + 6 months
  Single outcome measurement of body weight (kg).

SECONDARY OUTCOMES:
Change from baseline in metabolic status at 3 and 6 months | 0, + 3 months, + 6 months
  Composite outcome measure consisting of simultaneous measurment of: Glycaemia, Insulinemia, Homa index, Glycated Haemoglobin, Total Cholesterol, LDL cholesterol, HDL cholesterol, Triglyceredes; the composite outcome measured at 3 and 6 months.
Evaluation of immunological profile at baseline 3 and 6 months. | 0, + 3 months, + 6 months
  Composite outcome measure consisting of simultaneous measurment of: Full Count Blood Cell, ESR, Fibrinogen, Immunoglobulin, PCR; measured at baseline, 3 and 6 months.
Evaluation of bone deposition and resorption markers from baseline at 6 months | 0, + 6 months
  Composite outcome measure consisting of simultaneous measurment of: serum calcium, phosphate, parathyroid hormone (PTH), 25OH-vitamin D, phosphate, osteocalcin, bone phosphate alkaline (sBALP), serum-cross-linked N and C-telopeptide of bone type I collagen (NTx- CTx); measure at baseline and 6 months.
Evaluation of epicardial fat thickness from baseline at 6 months | 0, + 6 months
  Measurement of epicardial fat thickness (EFT) by hihg-resolution M-B-mode transthoracic echocardiography from baseline at 6 months.
Evaluation of hepatic steatosis from baseline at 6 months | 0, + 6 months
  Evaluation of hepatic steatosis by conventional ultrasound of the liver and with ASQ software with dedicated equipment and 7-5 Mhz convex probe frome baseline at 6 months.
Changes in quality of life from baseline at 2, 3 and 6 months | 0, + 2 months, +3 months, + 6 months
  Quality of life will be measured by questionnaires: AddiQol, Middle Sex Hospital Questionnaire (MHQ), International Index of Erectile Function (IIEF), Female Sexual Function Index (FSFI), Beck Depression Inventory Test (BDI-II).
Bone mineral density | 0, + 6 months
  Bone mineral density quantified by Dual X-Ray Absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — Dept. Experimental Medicine
Locations (1):
- Department of Experimental Medicine, Rome, Italy

REFERENCES:
- [Result] Nilsson AG, Marelli C, Fitts D, Bergthorsdottir R, Burman P, Dahlqvist P, Ekman B, Engstrom BE, Olsson T, Ragnarsson O, Ryberg M, Wahlberg J, Lennernas H, Skrtic S, Johannsson G. Prospective evaluation of long-term safety of dual-release hydrocortisone replacement administered once daily in patients with adrenal insufficiency. Eur J Endocrinol. 2014 Sep;171(3):369-77. doi: 10.1530/EJE-14-0327. Epub 2014 Jun 18. PMID 24944332
- [Result] Johannsson G, Nilsson AG, Bergthorsdottir R, Burman P, Dahlqvist P, Ekman B, Engstrom BE, Olsson T, Ragnarsson O, Ryberg M, Wahlberg J, Biller BM, Monson JP, Stewart PM, Lennernas H, Skrtic S. Improved cortisol exposure-time profile and outcome in patients with adrenal insufficiency: a prospective randomized trial of a novel hydrocortisone dual-release formulation. J Clin Endocrinol Metab. 2012 Feb;97(2):473-81. doi: 10.1210/jc.2011-1926. Epub 2011 Nov 23. PMID 22112807
- [Result] Johannsson G, Bergthorsdottir R, Nilsson AG, Lennernas H, Hedner T, Skrtic S. Improving glucocorticoid replacement therapy using a novel modified-release hydrocortisone tablet: a pharmacokinetic study. Eur J Endocrinol. 2009 Jul;161(1):119-30. doi: 10.1530/EJE-09-0170. Epub 2009 Apr 21. PMID 19383806
- [Derived] Venneri MA, Hasenmajer V, Fiore D, Sbardella E, Pofi R, Graziadio C, Gianfrilli D, Pivonello C, Negri M, Naro F, Grossman AB, Lenzi A, Pivonello R, Isidori AM. Circadian Rhythm of Glucocorticoid Administration Entrains Clock Genes in Immune Cells: A DREAM Trial Ancillary Study. J Clin Endocrinol Metab. 2018 Aug 1;103(8):2998-3009. doi: 10.1210/jc.2018-00346. PMID 29846607
- [Derived] Isidori AM, Venneri MA, Graziadio C, Simeoli C, Fiore D, Hasenmajer V, Sbardella E, Gianfrilli D, Pozza C, Pasqualetti P, Morrone S, Santoni A, Naro F, Colao A, Pivonello R, Lenzi A. Effect of once-daily, modified-release hydrocortisone versus standard glucocorticoid therapy on metabolism and innate immunity in patients with adrenal insufficiency (DREAM): a single-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Mar;6(3):173-185. doi: 10.1016/S2213-8587(17)30398-4. Epub 2017 Dec 8. PMID 29229498